CLINICAL TRIAL: NCT05801523
Title: Laparoscopic Therapy of Endometrioma: Sclerotherapy vs Cystectomy in Patients With Unfinished Reproductive Plans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Collaborators: University Hospital Ostrava (Other)
Responsible Party: Principal Investigator, Katarina Ivankova, Medical doctor at Endometriosis centre, Institute for the mother and child care, Institute for the Care of Mother and Child, Prague, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMHstudy
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Endometrioma; Endometriosis
Keywords: laparoscopic; sclerotherapy; endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic ethanol sclerotherapy (Active Comparator)
  Interventions: Procedure: laparoscopic ethanol sclerotherapy
- laparoscopic cystectomy (Active Comparator)
  Interventions: Procedure: laparoscopic cystectomy of endometrioma

INTERVENTIONS:
Procedure: laparoscopic ethanol sclerotherapy — ethanol (96%) sclerapy of endometrioma - endometrioma is filled with ethanol via foley catether, left for 10 min and than aspirated, endometrioma is washed with saline
  Arms: laparoscopic ethanol sclerotherapy
Procedure: laparoscopic cystectomy of endometrioma — cystectomy of endometrioma - removal of endometrioma from ovary surgically
  Arms: laparoscopic cystectomy

SUMMARY:
The aim of this prospective randomized study is to compare laparoscopic sclerotherapy to cystectomy in following: AMH dynamics, endometrioma recurrence, complications, pregnancy rate, assisted reproduction methods success rate, live birth rate

DETAILED DESCRIPTION:
Only patients who sign informed consent will be included. Only patients wishing for future pregnancy will be involved in the study. Expected number of enrolled subjects is 160 ( 80 in each arm) Patients with endometrioma and planned surgery to remove it will be randomized either to laparoscopic sclerotherapy with 96% ethanol or cystectomy. First AMH sample will be taken day before surgery. If other endometriosis lesions (deep or superficial) are present, they may be also resected during this surgery.

Ethanol sclerotherapy description: classical laparoscopic approach - small (max1cm) fenestration of endometrioma - aspiration of endometrioma contents- foley catheter insertion- ballon inflation inside of the cyst- instillation with 96% ethanol which is left in the cyst for 10min- aspiration of ethanol and flushing with saline.

Cystectomy: classical laparoscopic approach- large fenestration of endometrioma - aspiration of endometrioma contents- indentification of ovary/ endometrioma tissue and plane between the ovarian capsule and cyst wall is developed using a mix of blunt and sharp dissection - if bleeding is present it is stopped by cautious bipolar coagulation

visit 1 - surgery time (AMH day before surgery, age, BMI, endometriosis extent, gravidity/ parity, endometriosis residue after surgery, pain levels) visit 2- 3 months after surgery : Ultrasound, complications, pregnancy, asissted reproduction, pain levels visit 3+4 - 6/12months after surgery: AMH, Ultrasound, complications, pregnancy, asissted reproduction, pain levels visit 5- 24 months after surgery: Ultrasound, complications, pregnancy, asissted reproduction, pain levels

ELIGIBILITY:
Inclusion Criteria:

* IOTA benign endometrioma
* bilateral or unilateral endometrioma measuring 30 or more milimeters
* patients with unfinished reproductive plans

Exclusion Criteria:

* bilateral recurrence of endometrioma
* recurrent endometrioma if the other ovary is not present or patient had cystectomy on the other ovary
* suspision for ovarian malignancy
* signs of inflammatory pelvic disease
* disagreement with participation in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
AMH dynamics | Measuring change in AMH levels immediately before surgery and than at 6 and 12 months after surgery
  Measuring AMH level in blood
endometrioma recurrence | Measuring change of endometrioma size (in case of recurrence) at 3, 6, 12 and 24 months after surgery
  recurrence described as endometrioma measuring 20 or more milimeters on ultrasound
complications | 0-12 months
  recording all complications related to surgery, classified according Clavien Dindo

SECONDARY OUTCOMES:
Asissted reproduction methods succes rate | 0-24 months after surgery
  if patient undergoes assisted reproduction techniques and gets pregnant we check what methodes were used
pregnancy rate | 0-24 months after surgery
  pregnancy rate among study patients
deliveries | 24 months
  number of deliveries after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katarína Ivánková, MUDr., Principal Investigator — Institute for the Care of Mother and Child, Prague, Czech Republic
Locations (1):
- Institute for mother and child care, Prague, Czechia

REFERENCES:
- [Background] Falcone T, Flyckt R. Clinical Management of Endometriosis. Obstet Gynecol. 2018 Mar;131(3):557-571. doi: 10.1097/AOG.0000000000002469. PMID 29420391
- [Background] Busacca M, Vignali M. Ovarian endometriosis: from pathogenesis to surgical treatment. Curr Opin Obstet Gynecol. 2003 Aug;15(4):321-6. doi: 10.1097/01.gco.0000084247.09900.4f. PMID 12858105
- [Background] Cohen A, Almog B, Tulandi T. Sclerotherapy in the management of ovarian endometrioma: systematic review and meta-analysis. Fertil Steril. 2017 Jul;108(1):117-124.e5. doi: 10.1016/j.fertnstert.2017.05.015. Epub 2017 Jun 1. PMID 28579409
- [Background] Kasapoglu I, Ata B, Uyaniklar O, Seyhan A, Orhan A, Yildiz Oguz S, Uncu G. Endometrioma-related reduction in ovarian reserve (ERROR): a prospective longitudinal study. Fertil Steril. 2018 Jul 1;110(1):122-127. doi: 10.1016/j.fertnstert.2018.03.015. Epub 2018 Jun 20. PMID 29935810
- [Background] Crestani A, Merlot B, Dennis T, Chanavaz-Lacheray I, Roman H. Impact of Laparoscopic Sclerotherapy for Ovarian Endometriomas on Ovarian Reserve. J Minim Invasive Gynecol. 2023 Jan;30(1):32-38. doi: 10.1016/j.jmig.2022.10.001. Epub 2022 Oct 10. PMID 36228863
- [Background] De Cicco Nardone A, Carfagna P, De Cicco Nardone C, Scambia G, Marana R, De Cicco Nardone F. Laparoscopic Ethanol Sclerotherapy for Ovarian Endometriomas: Preliminary Results. J Minim Invasive Gynecol. 2020 Sep-Oct;27(6):1331-1336. doi: 10.1016/j.jmig.2019.09.792. Epub 2020 May 5. PMID 32380241
- [Background] Benaglia L, Somigliana E, Vercellini P, Abbiati A, Ragni G, Fedele L. Endometriotic ovarian cysts negatively affect the rate of spontaneous ovulation. Hum Reprod. 2009 Sep;24(9):2183-6. doi: 10.1093/humrep/dep202. Epub 2009 Jun 5. PMID 19502358
- [Background] Benaglia L, Somigliana E, Vighi V, Ragni G, Vercellini P, Fedele L. Rate of severe ovarian damage following surgery for endometriomas. Hum Reprod. 2010 Mar;25(3):678-82. doi: 10.1093/humrep/dep464. Epub 2010 Jan 17. PMID 20083485
- [Background] Jee BC. Efficacy of ablation and sclerotherapy for the management of ovarian endometrioma: A narrative review. Clin Exp Reprod Med. 2022 Jun;49(2):76-86. doi: 10.5653/cerm.2021.05183. Epub 2022 May 4. PMID 35698769
- [Background] Giampaolino P, Bifulco G, Di Spiezio Sardo A, Mercorio A, Bruzzese D, Di Carlo C. Endometrioma size is a relevant factor in selection of the most appropriate surgical technique: a prospective randomized preliminary study. Eur J Obstet Gynecol Reprod Biol. 2015 Dec;195:88-93. doi: 10.1016/j.ejogrb.2015.09.046. Epub 2015 Oct 24. PMID 26492167
- [Background] Garcia-Tejedor A, Martinez-Garcia JM, Candas B, Suarez E, Manalich L, Gomez M, Merino E, Castellarnau M, Regueiro P, Carreras M, Martinez-Franco E, Carrarrach M, Subirats N, Barbera J, Gonzalez S, Climent M, Fernandez-Montoli E, Ponce J. Ethanol Sclerotherapy versus Laparoscopic Surgery for Endometrioma Treatment: A Prospective, Multicenter, Cohort Pilot Study. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1133-1140. doi: 10.1016/j.jmig.2019.08.036. Epub 2020 Apr 7. PMID 32272240
- [Background] Aflatoonian A, Tabibnejad N. Aspiration versus retention ultrasound-guided ethanol sclerotherapy for treating endometrioma: A retrospective cross-sectional study. Int J Reprod Biomed. 2020 Nov 22;18(11):935-942. doi: 10.18502/ijrm.v13i11.7960. eCollection 2020 Nov. PMID 33349801